CLINICAL TRIAL: NCT04216108
Title: Comparative Study 23G Versus 27G Vitrectomy
Acronym: 23Gvs27G
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Peter Stalmans (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Peter Stalmans, Prof. Dr. Peter Stalmans, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S61408
Record Dates: First submitted 2019-07-15; First posted 2020-01-02 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Vitreoretinal Surgery
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 23G gauge needle vitrectomy surgery (Experimental)
  Interventions: Device: Vitrectomy (23G gauge needle)
- 27G gauge needle vitrectomy surgery (Experimental)
  Interventions: Device: Vitrectomy (27G gauge needle)

INTERVENTIONS:
Device: Vitrectomy (23G gauge needle) — Vitrectomy surgery with 23G gauge needle technique
  Arms: 23G gauge needle vitrectomy surgery
Device: Vitrectomy (27G gauge needle) — Vitrectomy surgery with 27G gauge needle technique
  Arms: 27G gauge needle vitrectomy surgery

SUMMARY:
Investigator-initiated, comparative double-arm, mono-center, prospective, interventional case study to determine whether ultra-small gauge surgery (27G gauge needle) improves postoperative outcome and patient morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18
* No prior vitrectomy surgery in the study eye
* No prior inclusion in this trial
* Scheduled for vitrectomy for floater removal or macular surgery

Exclusion Criteria:

* Patients with serious heart, lung, liver, or kidney dysfunction
* Patients with proliferative diabetic retinopathy, endophthalmitis, uveitis and other eye disease that impacts the outcome of vitrectomy surgery Patients with HIV (Human Immune-deficiency Virus)
* Patients with history of drug abuse or alcoholism
* Patients participating in other drug or medical device clinical trials before screening for this trial
* Pregnancy, preparation for pregnancy during clinical trial, or breastfeeding
* Belief by the investigator that a patient's condition would hinder the clinical trial, such as a patient prone to mental stress, loss of control of mood, or depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Changes in post-operative outcome of pain | 1 week
  By assessing the amount of pain on a visual analogue scale (score 0 - 9)
Changes in post-operative outcome of redness | 1 week
  Scoring the amount of redness on a scale 0-4 through eye photos
Changes in post-operative outcome of measured inflammation | 1 week
  Measuring the amount of inflammation by measurement of Flare (photon/ms)
Changes in post-operative outcome in grading of anterior chamber cells | 1 week
  Clinical assesment by slit lamp (Tyndall 0 - 3 and Cells 0 - 3)

SECONDARY OUTCOMES:
Post-operative parameter: Visual acuity | 1 week
  Best corrected visual acuity in LogMar will be obtained to report the visual acuity.
Post-operative parameter: Intraocular pressure | 1 week
  Millimeter of Mercury pressure (mmHG) will be measured to report the intraocular pressure.
Post-operative parameter: Pain assessment | 1 week
  A questionnaire with visual analogue scale will be used to assess the level of pain up to 1 week after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stalmans, MD Phd, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven (UZ Leuven), Leuven, Vl-Brabant, Belgium